CLINICAL TRIAL: NCT04372550
Title: Pathophysiological Mechanisms and Early Exercise Rehabilitation Counter Measures of Hypermetabolism and Muscle Wasting in Severe Burns.
Brief Title: Effects of Early Exercise Rehabilitation in Severe Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Research Foundation Flanders (Other); Wuhan Third Hospital (Other)
Responsible Party: Principal Investigator, Ulrike Van Daele, Prof. dr., Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11B8619N
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Burns
Keywords: Burns; Exercise rehabilitation; Exercise Therapy; Muscle wasting; Hypermetabolism; Insulin resistance
MeSH Terms: conditions — Burns; Muscular Atrophy; Insulin Resistance | interventions — Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Masking Description: Analysis of the primary outcome is carried out blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care treatment:
  - including passive / assisted / active movements, stretching, functional exercise, scar treatment
  Duration: 6-12 weeks
  Interventions: Other: Standard of Care
- Exercise (Experimental): Standard of care + added exercises
  Exercise type: resistance and aerobic exercise
  Resistance Exercise: 3x / week (manual resistance, free weights, machines) Aerobic exercise: 2x / week (cycle ergometer, treadmill)
  Duration: 6-12 weeks
  Interventions: Other: Exercise; Other: Standard of Care

INTERVENTIONS:
Other: Exercise — Resistance and aerobic exercise in addition to standard of care rehabilitation
  Arms: Exercise
Other: Standard of Care — Standard of care rehabilitation

SUMMARY:
BACKGROUND:

Postburn changes in glucose and protein metabolism are at their peak during the acute phase of severe burns. The resulting metabolic derangements lead to substantial muscle wasting, insulin resistance, which ultimately hampers full recovery and reintegration into society.

PURPOSE:

This randomized controlled trial was initiated to investigate the effects of exercise-based rehabilitation on muscle wasting, insulin resistance, and quality of life during the acute phase of severe adult burns.

METHODS:

Severly burned adults (40-80%TBSA) will be recruited from one of China's largest burn centres.

Subjects allocated to the intervention group will undergo a 6-12 week long exercise program in addition to standard care rehabilitation. As part of the exercise program, participants will carry out progressive resistance and aerobic training, initiated as soon as medical safety and patient cooperation allow. Exercise type and dosage will be chosen according to patient status in terms of grafts, mobility, and strength.

The control group will receive standard care rehabilitation only, including passive, assisted, active range of motion exercise, functional exercise, and scar treatment.

The results of this translational research will provide insight into the effects and mechanisms of exercise on both a fundamental and clinical spectrum.

DETAILED DESCRIPTION:
The added exercise intervention is initiated in line with the following readiness criteria, which were checked prior to each training session:

Criteria:

* Cardiorespiratory stability:
* Mean arterial pressure (MAP) 60 - 110 mmHg
* fraction of inspired oxygen (FiO2) <60%
* partial pressure of oxygen / fraction of inspired oxygen (PaO2/FiO2) >200
* Respiratory rate <40 bpm
* Positive end expiratory pressure (PEEP) <10 cmH2O
* no high inotropic doses (Dopamine >10 mcg/kg/min or Nor/adrenaline <0,1 mcg/kg/min)
* Temp. 36 - 38,5°C
* Richmond Agitation Sedation Scale (RASS) -2 - +2
* Medical Doctor clearance
* Medical research council (MRC) score lower limbs ≥3

Accordingly, the post burn starting time differs per enrolled subject.

Exercises are administered as in-bed exercises or out-of-bed exercises, depending on whether subjects are able and allowed to engage in out-of-bed mobility.

Exercise intensity for resistance training is set at 60% peak force based on a weekly peak force measurement by hand-held dynamometry, or on a 3 RM in case of out of bed exercises. Aerobic exercise intensity is set at 50-75% peak Watts determined by a weekly cycle ergometer or treadmill ramp protocol.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 - ≤70 %TBSA
* Burn depth: 2nd deep / 3rd degree

Exclusion Criteria:

* Electrical burn (except flash burns)
* Associated injury: fracture lower limb
* Diabetes Mellitus type 1
* Central neurological/neuromuscular disorders (interfering with assessment/exercise)
* Cognitive / psychological disorders (interfering with cooperation)
* Cardiopulmonary disease (interfering with exercise safety)
* Pregnancy
* Palliative care

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in quadriceps muscle layer thickness (QMLT) | Baseline - 12 weeks
  Method: B-mode ultrasound on the anterior aspect of the thigh. Technique: maximal and minimal pressure Location: measured at 1/2 and 2/3 of the distance between anterior superior iliac spine and the superior pole of the patella.
  Analysis: An average of 3 trials will be recorded and analyzed using dedicated software
Change in rectus femoris cross sectional area (RF-CSA) | Baseline - 12 weeks
  Method: B-mode ultrasound on the anterior aspect of the thigh. Technique: minimal pressure. Location: measured at the most proximal distance where the entire muscle belly is still visible on the ultrasound image.
  Analysis: An average of 3 trials will be recorded and analyzed using dedicated software.

SECONDARY OUTCOMES:
Change in insulin resistance | Baseline and 12 weeks
  Method: HOMA-2 calculated by fasting plasma glucose and insulin, analysed by Western Blot Chemiluminescence

OTHER OUTCOMES:
Change in Interleukin-1 | Baseline and 12 weeks
  Western Blot Chemiluminescence
Change in Interleukin-6 | Baseline and 12 weeks
  Western Blot Chemiluminescence
Change in Tumor Necrosis Factor alpha (TNF-α) | Baseline and 12 weeks
  Western Blot Chemiluminescence
Change in C-reactive protein | Baseline and 12 weeks
  Western Blot Chemiluminescence
Change in Insulin like growth factor 1 (IGF-1) | Baseline and 12 weeks
  Western Blot Chemiluminescence
Change in Glucagon | Baseline and 12 weeks
  ELISA kits DGCG0, R&D Systems, Inc, USA
Change in Myostatin | Baseline and 12 weeks
  ELISA kits DGDF80, R&D Systems, Inc, USA
Change in isometric peak force (knee extension) | Baseline and 12 weeks
  Method: Hand-held dynamometry (Lafayette instrument Co. Europe, U.K.). Isometric peak fore is measured by a 'make' manoeuvre with a fixation band disallowing movement.
  Test position: Supine with a fixation band fixed to the hospital bed. Analysis: Best of 3 trials
Change in isometric peak force (hip flexion) | Baseline and 12 weeks
  Method: Hand-held dynamometry (Lafayette instrument Co. Europe, U.K.). Isometric peak fore is measured by a 'make' manoeuvre with a fixation band disallowing movement.
  Test position: Supine with a fixation band fixed to the hospital bed. Analysis: Best of 3 trials
Change in isometric peak force (hip extension) | Baseline and 12 weeks
  Method: Hand-held dynamometry (Lafayette instrument Co. Europe, U.K.). Isometric peak fore is measured by a 'make' manoeuvre with a fixation band disallowing movement.
  Test position: Supine with a fixation band fixed to the hospital bed. Analysis: Best of 3 trials
Change in hand grip strength | Baseline and 12 weeks
  Method: Baseline LITE hydraulic dynamometer Analysis: Best of 3 trials
Change in Burn Specific Health Scale-Brief (BSHS-B) | Baseline and 12 weeks
  Burn-specific quality of life, measured by the Burn Specific Health Scale-Brief questionnaire (Mandarin Chinese version).
  Total score 152 (0 worst score, 152 best score), consisting of 6 subdomains:
  1) Body imagine (36 points) Simple abilities (36 points) Sexuality (24 points) Affect (32 points) Work (16 points) Interpersonal relationship (8 points)
Change in EQ-5D-5L | Baseline and 12 weeks
  Overall quality of life, measured by EQ-5D-5L (Mandarin Chinese version) Total score: 25 points (0 worst score, 25 best score), consisting of 5 subdomains
  1. Mobility (5 points)
  2. Self-care (5 points)
  3. Usual activities (5 points)
  4. pain / discomfort (5 points)
  5. Anxiety / Depression (5 points) EQ overall health assessed on a Visual Analogue Scale, Total 0-100 (0 worst, 100 best score)
Number of adverse events | Baseline and 12 weeks
  Recording of complications during exercise: Graft take, Wound infections, Medical, Cardio-respiratory safety

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Van Daele, Principal Investigator — Faculty of Medicine and Health Sciences, University of Antwerp
Locations (1):
- Institute of Burns, Wuhan Third Hospital & Tongren Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Datasets will be made available upon request.